CLINICAL TRIAL: NCT04705090
Title: A Single-arm, Open, Multicenter, Phase II Study to Investigate the Efficacy and Safety of YY-20394 in Patients With Relapsed or Refractory Peripheral T/NK Cell Lymphoma
Brief Title: A Study of YY-20394 in Patients With Relapsed or Refractory Peripheral T/NK Cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai YingLi Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YY-20394-010
Record Dates: First submitted 2021-01-08; First posted 2021-01-12 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2020-12

CONDITIONS: PTCL

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- YY-20394 treatment (Experimental): YY-20394 tablets, 20mg spec, 80mg QD, 28 days for each cycle.
  Interventions: Drug: YY-20394 treatment

INTERVENTIONS:
Drug: YY-20394 treatment — Each treatment cycle is comprised of 28-day consecutive dosing of YY-20394, 80mg QD (days 1 to 28). Upon completion of each cycle, patients may continue to receive oral YY-20394 tablets if they are benefit from the treatment and the toxicity is tolerable.

SUMMARY:
A single-arm, open, multicenter study to investigate the efficacy and safety of YY-20394, an oral small molecular inhibitor of PI3K-delta, in patients with relapsed or refractory peripheral T/NK cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Males and/or females over age 18.
* Histologically or cytologically confirmed diagnosis of relapsed or refractory peripheral T/NK cell lymphoma.
* Eastern Cooperative Oncology Group performance status of 0 to 1.
* Life expectancy of at least 3 months.
* At least one measurable lesion according to Lugano 2014.
* Adequate organ function.
* Had anti-tumor treatment within 2 weeks prior to the first dose of investigational product (including TKI, Chinese herbal anti-tumor treatment); within 4 weeks prior to the first dose of investigational product (including chemotherapy, radiotherapy, immunotherapy and major surgery); other targeted therapies with 5 half-life period prior to the first dose.
* Men and women of childbearing potential are willing to employ an effective method of contraception for the entire duration of study and 6 months after the last dose.
* Volunteers did not participate in other clinical trials within 1 month prior to study entry.
* Provision of signed and dated, written informed consent prior to any study- specific evaluation.

Exclusion Criteria:

* Previous treatment with any PI3K-delta inhibitors.
* Uncontrolled pleural effusion and ascites.
* The dosage of steroid hormone (prednisone equivalent) was greater than 20mg/day, and lasted for more than 14 days.
* Medical conditions in swallowing difficulty, malabsorption, or other chronic gastrointestinal disease that may hamper compliance and/ or absorption of the investigational agent.
* Drugs that may prolong the QT (such as anti-arrhythmic drugs) could not be interrupted during the study period.
* Evidence of central nervous system involvement of the malignancy, including invasion of brain parenchyma and meninges, or spinal cord compression.
* Have active viral, bacterial, fungal, or other infections that require systematic treatment (e.g., active tuberculosis), excluding nail bed fungal infections.
* Active infection with hepatitis B and C virus (volunteers with HBsAg or HBcAb positive but HBV-DNA negative, or HCV antibody positive but HCV-RNA negative can be enrolled).
* History of immune deficiency (acquired and congenital), or history of organ transplantation, or allogeneic bone marrow or hematopoietic stem cell transplantation; with active autoimmune disease or history of autoimmune disease (e.g., autoimmune enteritis and systemic lupus erythematosus).
* prior autologous hematopoietic stem cell transplantation within 90 days prior to the first dose of study drug.
* Presence of severe or uncontrolled cardiovascular disease.
* Medical history of active bleeding within 2 months prior to study entry, or currently achieved anticoagulant therapy, or susceptible to bleed by the judgement of investigator.
* Presence of concomitant diseases that are seriously endanger the safety of patient or affect the completion of the study by the investigator's judgment (e.g., uncontrolled hypertension, diabetes, thyroid diseases).
* Had received GCSF or blood transfusion treatment within 14 days prior to study entry.
* Female subjects of childbearing potential have a positive pregnancy test at the baseline.
* Medical history of other primary malignant tumors in the past 5 years except for the following: clinically cured cervical or breast carcinoma in situ, local basal cell or squamous cell carcinoma of the skin, thyroid tumor.
* Adverse events occurred during previous anticancer therapy have not been recovered to ≤1 (CTCAE 5.0) except toxicity with no significant risk determined by investigator such as alopecia.
* Live vaccine was administered within 30 days prior to the first dose of the investigational drug, or was scheduled to be administered during the study period.
* Judgment by the investigator that the volunteer should not participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-04 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
ORR | up to 12 months
  Objective Response Rate

SECONDARY OUTCOMES:
DOR | up to 12 months
  Duration of response
PFS | up to 12 months
  Progression free survival
DCR | up to 12 months
  Disease control rate
TTR | up to 12 months
  Time to response
Safety and Tolerability | up to 12 months
  safety and tolerability of investigational Product assessed as the number of participants experiencing adverse events (AEs, CTCAE5.0) or abnormalities in vital signs, laboratory tests, or electrocardiograms.

IPD SHARING:
Plan to Share IPD: No